CLINICAL TRIAL: NCT07184476
Title: Assessment of Microvascular Circulation in the Pediatric Cardiac Surgery Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sitaram Emani, Associate Professor of Surgery, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00050326
Record Dates: First submitted 2025-08-07; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Tetrology of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Tetrology of Fallot repair: Cyanotic physiology with Tetrology of Fallot w/pulmonary stenosis or atresia
- Primary ventricular septal defect repair (VSD): Acyanotic lesion with VSD repair patch graft

SUMMARY:
The pediatric cardiac surgery patient endures a tremendous number of physiologic alterations during surgery and cardiopulmonary bypass (CPB) that lasts well into the recovery period. Most of the hemodynamic data are assessed and treated with macrovascular assessment tools such as blood pressure and central venous line measures. Studies show there may be an incoherence of macrovascular to microvascular assessment; i.e. a patient with a stable macrovascular status may not be in the state of microvascular stability. The use of a handheld device called Cytocam incident dark-field (IDF) microcirculatory camera (Braedius Medical, Huizen, Netherlands) gives real-time video screening and data feedback to assess the microvasculature in the hemodynamically labile patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary diagnosis of ventricular septal defect or tetrology of Fallot

Exclusion Criteria:

* Critical airway, congenital genetic abnormality of the mouth/tongue

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be identified by preoperative assessment at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Braedius Cytocam efficacy in the pediatric surgery patient | - After intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB) initiated - after cross clamp placed - every hour on CPB - after CPB ends - every 4 hours during the first 48 hours after admitted to the intensive care unit
  Evaluate the effective use of handheld vital microscopy (HVM), i.e. the Cytocam incident dark-field (IDF) microvascular camera along with CCTools software (Braedius-Medical Huizen, The Netherlands) in the microvasculature for pediatric cardiac surgery patient.
Capillary density measurements | - After intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB)initiated - After cross clamp placed - every hour on CPB - after CPB ends - every 4 hours during the first 48 hours after admitted to the intensive care unit
  Evaluate perioperative microcirculatory changes with relationship to routine clinical interventions in pediatric cardiac surgery care: Perfused vessel density (PVD) mm squared x mm squared (both continuous and categorical: lowest quartile vs rest) assessed per CCTools software.
Microcirculatory flow index grading | - After intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB) initiated - after cross clamp placed - every hour on CPB - after CPB ends - every 4 hours during the first 48 hours after admitted to the intensive care unit
  Microcirculatory flow index (MFI) (both continuous - a qualitative score graded as having no flow, intermittent, sluggish, or continuous flow ranging from 0 (no flow) to 3 (normal flow) with < 2.6 defined as disturbed perfusion quality - categorical).
Surrogates of tissue perfusion and acute kidney injury | - After intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB) initiated - after cross clamp placed - every hour on CPB - after CPB ends - every 4 hours during the first 48 hours after admitted to the intensive care unit
  Surrogate of tissue perfusion with low urine output (<0.5ml/kg/hr > 1 yr, < 1 ml/kg/hr < 1 yr). Chi-squared and Correlation analysis

SECONDARY OUTCOMES:
Early outcome measures of prolonged ventilator times | - after intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB)initiated - after cross clamp placed - every hour on CPB - after CPB ends - every 4 hours during the first 48 hours after admitted to the intensive care unit
  Are microcirculatory changes associated with early outcome measures in pediatric patients? Association between microcirculation assessment of Perfused vessel density (PVD) mm squared x mm squared (both continuous and categorical: lowest quartile vs rest) assessed per CCTools software and prolonged ventilator times as defined by >48 hours.
Adverse outcomes | - after intubation in operation room - 10 minutes after cardiopulmonary bypass (CPB) initiated - after cross clamp placed - every hour on CPB - every 4 hours during the first 48 hour after admitted to the intensive care unit
  Are microcirculatory changes associated with adverse outcomes in pediatric patients? Association of microcirculation flow index <2.6 (no units - using the Massey grading system) with the semi-automatic software analysis (CCTools). Averaging the values of each time point to major adverse reaction of stroke

IPD SHARING:
Plan to Share IPD: Undecided
Determining efficacy of using the device in Boston Childrens Hospital

REFERENCES:
- [Background] Mukaida H, Matsushita S, Kuwaki K, Inotani T, Minami Y, Saigusa A, Amano A. Time-dose response of oxygen delivery during cardiopulmonary bypass predicts acute kidney injury. J Thorac Cardiovasc Surg. 2019 Aug;158(2):492-499. doi: 10.1016/j.jtcvs.2018.10.148. Epub 2018 Nov 16. PMID 30578056
- [Background] Favia I, Garisto C, Rossi E, Picardo S, Ricci Z. Fluid management in pediatric intensive care. Contrib Nephrol. 2010;164:217-226. doi: 10.1159/000313733. Epub 2010 Apr 20. PMID 20428006
- [Background] Massey MJ, Larochelle E, Najarro G, Karmacharla A, Arnold R, Trzeciak S, Angus DC, Shapiro NI. The microcirculation image quality score: development and preliminary evaluation of a proposed approach to grading quality of image acquisition for bedside videomicroscopy. J Crit Care. 2013 Dec;28(6):913-7. doi: 10.1016/j.jcrc.2013.06.015. Epub 2013 Aug 21. PMID 23972316
- [Background] Erdem O, de Graaff JC, Hilty MP, Kraemer US, de Liefde II, van Rosmalen J, Ince C, Tibboel D, Kuiper JW. Microcirculatory Monitoring in Children with Congenital Heart Disease Before and After Cardiac Surgery. J Cardiovasc Transl Res. 2023 Dec;16(6):1333-1342. doi: 10.1007/s12265-023-10407-4. Epub 2023 Jul 14. PMID 37450208
- [Background] Mendelson AA, Lam F, Peirce SM, Murfee WL. Clinical perspectives on the microcirculation. Microcirculation. 2021 Apr;28(3):e12688. doi: 10.1111/micc.12688. No abstract available. PMID 33629399
- [Background] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Background] Selewski DT, Cornell TT, Heung M, Troost JP, Ehrmann BJ, Lombel RM, Blatt NB, Luckritz K, Hieber S, Gajarski R, Kershaw DB, Shanley TP, Gipson DS. Validation of the KDIGO acute kidney injury criteria in a pediatric critical care population. Intensive Care Med. 2014 Oct;40(10):1481-8. doi: 10.1007/s00134-014-3391-8. Epub 2014 Jul 31. PMID 25079008
- [Background] Kuiper JW, Tibboel D, Ince C. The vulnerable microcirculation in the critically ill pediatric patient. Crit Care. 2016 Oct 30;20(1):352. doi: 10.1186/s13054-016-1496-x. PMID 27794361
- [Background] Top AP, Ince C, Schouwenberg PH, Tibboel D. Inhaled nitric oxide improves systemic microcirculation in infants with hypoxemic respiratory failure. Pediatr Crit Care Med. 2011 Nov;12(6):e271-4. doi: 10.1097/PCC.0b013e31820ac0b3. PMID 21297516
- [Background] Watchorn JC, Fargaly H, Gilani M, Assadi J, Deitchman AR, Naumann DN, Wollborn J, Goebel U, McCurdy MT, Hutchings SD. The Reproducibility of the Point of Care Microcirculation (POEM) Score When Used to Assess Critically Ill Patients: A Multicenter Prospective Observational Study. Shock. 2020 Jul;54(1):15-20. doi: 10.1097/SHK.0000000000001474. PMID 31764623
- [Background] Gilbert-Kawai E, Coppel J, Bountziouka V, Ince C, Martin D; Caudwell Xtreme Everest and Xtreme Everest 2 Research Groups. A comparison of the quality of image acquisition between the incident dark field and sidestream dark field video-microscopes. BMC Med Imaging. 2016 Jan 21;16:10. doi: 10.1186/s12880-015-0078-8. PMID 26797680
- [Background] Alten JA, Klugman D, Raymond TT, Cooper DS, Donohue JE, Zhang W, Pasquali SK, Gaies MG. Epidemiology and Outcomes of Cardiac Arrest in Pediatric Cardiac ICUs. Pediatr Crit Care Med. 2017 Oct;18(10):935-943. doi: 10.1097/PCC.0000000000001273. PMID 28737598
- [Background] Scolletta S, Marianello D, Isgro G, Dapoto A, Terranova V, Franchi F, Baryshnikova E, Carlucci C, Ranucci M. Microcirculatory changes in children undergoing cardiac surgery: a prospective observational study. Br J Anaesth. 2016 Aug;117(2):206-13. doi: 10.1093/bja/aew187. PMID 27440632
- [Background] Buijs EA, Verboom EM, Top AP, Andrinopoulou ER, Buysse CM, Ince C, Tibboel D. Early microcirculatory impairment during therapeutic hypothermia is associated with poor outcome in post-cardiac arrest children: a prospective observational cohort study. Resuscitation. 2014 Mar;85(3):397-404. doi: 10.1016/j.resuscitation.2013.10.024. Epub 2013 Nov 5. PMID 24200889
- [Background] Akin S, Dos Reis Miranda D, Caliskan K, Soliman OI, Guven G, Struijs A, van Thiel RJ, Jewbali LS, Lima A, Gommers D, Zijlstra F, Ince C. Functional evaluation of sublingual microcirculation indicates successful weaning from VA-ECMO in cardiogenic shock. Crit Care. 2017 Oct 26;21(1):265. doi: 10.1186/s13054-017-1855-2. PMID 29073930
- [Background] Aksu U, Yavuz-Aksu B, Goswami N. Microcirculation: Current Perspective in Diagnostics, Imaging, and Clinical Applications. J Clin Med. 2024 Nov 10;13(22):6762. doi: 10.3390/jcm13226762. PMID 39597906
- [Background] Hilty MP, Guerci P, Ince Y, Toraman F, Ince C. MicroTools enables automated quantification of capillary density and red blood cell velocity in handheld vital microscopy. Commun Biol. 2019 Jun 19;2:217. doi: 10.1038/s42003-019-0473-8. eCollection 2019. PMID 31240255
- [Background] Ince C, Boerma EC, Cecconi M, De Backer D, Shapiro NI, Duranteau J, Pinsky MR, Artigas A, Teboul JL, Reiss IKM, Aldecoa C, Hutchings SD, Donati A, Maggiorini M, Taccone FS, Hernandez G, Payen D, Tibboel D, Martin DS, Zarbock A, Monnet X, Dubin A, Bakker J, Vincent JL, Scheeren TWL; Cardiovascular Dynamics Section of the ESICM. Second consensus on the assessment of sublingual microcirculation in critically ill patients: results from a task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2018 Mar;44(3):281-299. doi: 10.1007/s00134-018-5070-7. Epub 2018 Feb 6. PMID 29411044
- [Background] Dilken O, Ergin B, Ince C. Assessment of sublingual microcirculation in critically ill patients: consensus and debate. Ann Transl Med. 2020 Jun;8(12):793. doi: 10.21037/atm.2020.03.222. PMID 32647718
- See also: Braedius Medical Cytocam Microcirculation camera website — https://www.braedius-medical.com/